CLINICAL TRIAL: NCT06286202
Title: Integrative Neuro-social Cognitive Strategy Programme for Instilling REcovery (INSPIRE): a Community-Based Cognitive Remediation Trial
Brief Title: Integrative Neuro-social Cognitive Strategy Programme for Instilling REcovery (INSPIRE) a Community-Based Cognitive Remediation Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Technology (Other)
Collaborators: Singapore Anglican Community Services (Unknown)
Responsible Party: Principal Investigator, Bhing-Leet Tan, Professor and Cluster Director, Singapore Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECAS-0306
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: cognitive remediation; Neuropsychological and Educational Approach to Remediation; Multicontext Treatment Approach; metamotivation; psychiatric rehabilitation; schizophrenia; community mental health
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: The intervention study model is a parallel randomized controlled trial. There will be two arms. The experimental arm is 'cognitive remediation' and the control arm is 'standard psychiatric rehabilitation'. Participants will be assigned to one of the treatment arms at the beginning of the trial and will continue in that arm throughout the length of the trial. Assignment to the group is done using a computer randomization generator. All eligible participants will be randomly assigned to one of the treatment arms (experimental or control arm) based on a 1:1 treatment allocation. Hence, those who are randomly allocated to the experimental arm will receive cognitive remediation throughout the trial, while those randomly allocated to the control arm will receive standard psychiatric rehabilitation throughout the trial. Both treatment arms will run in parallel.
Who Masked: Outcomes Assessor
Masking Description: Upon randomization, the co-investigators will indicate the allocated group in a separate spreadsheet from the outcome measurements. The co-investigator who is collecting baseline, post-intervention and 8-week outcome measurements will be blinded to the treatment allocation of each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Remediation: Adapted Neuropsychological and Education Approach to Remediation (NEAR) (Experimental): NEAR consists of using carefully selected computer cognitive games to restore cognitive functioning through rehearsal and strategy learning. It will be delivered 3 times a week for 12 weeks at the center. The duration of each session within the week is as follows: 1) First session: 45 min computer-assisted cognitive exercises + 30 min bridging group; 2) Second session: 30 min computer-assisted cognitive exercises + 45 min bridging group; 3) Third session: 45 min computer-assisted cognitive exercises. Computer-assisted cognitive exercises are sessions where participants engage in cognitive games that target different cognitive domains. In addition, the Multicontext Treatment Approach to strategy learning will be carried out. The metacognitive framework of self-evaluation and activity mediation will also be utilized. Bridging groups are conducted twice a week, to aid transfer of learning from the computer game sessions to the participants' everyday life.
  Interventions: Behavioral: Cognitive Remediation: Adapted Neuropsychological and Education Approach to Remediation (NEAR)
- Standard Psychiatric Rehabilitation at Anglican Care Centers (Other): Participants in the control arm will attend their scheduled activities at their respective Anglican Care Centers. The Anglican Care Centers run a variety of activities to provide psychosocial rehabilitation for clients with serious mental illness. These may include vocational training such as training in a retail shop or café, instrumental activities of daily living training (eg: taking public transport, money management), psychoeducation, social skills training etc. Participants in the control arm will not be enrolled into the cognitive remediation.
  Interventions: Behavioral: Standard Psychiatric Rehabilitation at Anglican Care Centers

INTERVENTIONS:
Behavioral: Cognitive Remediation: Adapted Neuropsychological and Education Approach to Remediation (NEAR) — NEAR consists of computer-assisted cognitive exercises to restore cognitive functioning through rehearsal and strategy learning. Based on the results of the baseline assessments, the therapist will complete the Cognitive Remediation Treatment Plan, to outline targeted cognitive domains and functional goals. During the cognitive games sessions, the Multicontext Treatment Approach will be used, where error patterns are identified. The participants will work on metacognition and use of strategies to overcome challenges faced during the computer games sessions. Bridging groups may include activities for participants to utilize strategies learnt during the computer game sessions to everyday living. Participants will also learn about cognitive impairments and how lifestyle modifications, mood regulation etc can affect cognitive performance. In addition, they will learn about metamotivation and build awareness about their motivation levels through self- reflection and self-monitoring.
  Arms: Cognitive Remediation: Adapted Neuropsychological and Education Approach to Remediation (NEAR)
Behavioral: Standard Psychiatric Rehabilitation at Anglican Care Centers — Participants in the control arm will attend their usual psychiatric rehabilitation activities. These activities may include vocational training, community living skills training, psychoeducation, social skills training and peer support etc. These activities are also undertaken by participants in the experimental arm.
  Arms: Standard Psychiatric Rehabilitation at Anglican Care Centers

SUMMARY:
Adults with serious mental illnesses (such as schizophrenia and schizoaffective disorders) often experience a range of cognitive difficulties (such as memory, problem solving difficulties) that affect their ability to lead meaningful life roles. Cognitive remediation is an intervention to address cognitive difficulties in this group of mental health service users. Its implementation in less well-resourced community-based settings is less well-studied.

Therefore, the aims of the study are:

* To investigate the effects of cognitive remediation on various cognitive skills (such as attention, memory, problem-solving, facial expression recognition, taking others' perspectives etc), for participants with schizophrenia or schizoaffective disorders in community mental health settings.
* To investigate if factors such as participants' motivation for engagement and social interaction can affect changes in cognitive skills and functional ability.

Participants in the treatment group will attend computer-based cognitive exercises to improve their cognitive skills. They will also participate in group sessions facilitated by therapists to learn how to utilize strategies learned from the computer sessions in their daily lives. Participants in the control group will attend the usual rehabilitation activities in their respective community-based psychiatric rehabilitation centers.

This research study will compare the differences in their cognitive performance, functional ability and recovery immediately after the intervention and 8 weeks later.

DETAILED DESCRIPTION:
Persons with severe mental illness such as schizophrenia and schizoaffective disorders often have difficulties integrating back to the community and many face the prospect of long-term institutionalisation when families could not manage them. It is assumed that their inability to function is due to their mood and psychotic symptoms such as auditory hallucinations and persecutory delusions and paranoid thoughts. However, evidence has shown that neurocognitive impairment (such as information processing, memory, problem solving) coupled with social cognitive problems (such as difficulty with emotion recognition, perspective taking etc) are the ones with more long-term impact on their functioning (Green et.al., 2000; Tan, 2009).

Cognitive remediation is a form of intervention that addresses cognitive impairments of persons with psychiatric conditions, in order to improve real-world functioning. There are several approaches to cognitive remediation. One of the well-studied cognitive remediation programmes is the Neuropsychological and Educational Approach to Remediation (NEAR), which consists of computer-assisted cognitive exercises, followed by bridging sessions to generalise strategies learnt to daily living. NEAR is conducted in groups of 5-8 clients and is facilitated by 1-2 therapists (Medalia, Revheim and Herlands, 2009). It uses drill-and-practice rehearsal method to improve discrete cognitive skills, as well as strategy-learning method to equip clients with strategies to overcome cognitive challenges in different functional scenarios. NEAR has been implemented in inpatient wards, supported housing settings and outpatient rehabilitation settings in United States and other countries, largely with schizophrenia and schizoaffective disorders clients (Medalia et.al., 2000, 2003, 2019). In Singapore, cognitive remediation has been conducted in early psychosis intervention service with positive results (Chong et.al., 2021).

Meta-analyses of cognitive remediation has shown that while the rehearsal approach improves cognitive performance, the strategy learning approach has a greater effect size on functional outcomes (McGurk et.al., 2007; Wykes et.al., 2011). Deepening strategy learning in cognitive remediation is thus an important ingredient within cognitive remediation. In occupational therapy practice, the Multicontext Treatment Approach has been established as a credible and evidence-based framework on strategy learning (Toglia et.al, 2011, 2020). It utilises an over-arching metacognitive strategy approach that focuses on promoting self-awareness, self-monitoring skills, strategy generation and effective strategy use across a wide range of functional activities. The therapist works closely with the service user to determine single or multiple strategies that can be applied across a broad range of occupations, activities and tasks (Toglia, 2018). Thus, incorporating the Multicontext Treatment Approach as a strategy learning framework within NEAR will enhance skills acquisition for persons with cognitive impairment and may yield better functional outcomes.

In addition, literature over the past decade has highlighted the overlapping constructs between neurocognition, social cognition and negative symptoms in the pathway between symptomatology and functional outcomes (Hajdúk, et.al., 2021; Ventura et.al., 2009). Therefore, integrated neuro and social cognitive remediation have been developed, with some positive findings (DeMare et.al., 2019; Tan et.al., 2018) Such interventions, when contextualised to service users' occupational context, have been shown to improve social functioning and community independence (Mueller et.al., 2015. Furthermore, negative symptoms such as low motivation (ie: avolition) appears to play a significant mediating role in the outcomes of cognitive remediation (Lynch et.al., 2022). Therefore, strategies to enhance motivation, specifically the self-awareness and monitoring of motivation (ie: metamotivation) have also been considered as part of strategy learning.

In light of recent advancement in the research of cognitive remediation, this study attempts to integrate current knowledge in the various therapeutic ingredients of cognitive remediation to deliver an adapted NEAR intervention that meets the needs of community-dwelling persons with schizophrenia and schizoaffective disorders. The adapted NEAR intervention, which comprises of computer-based cognitive exercises and bridging groups, will be implemented in five community psychiatric rehabilitation centers, namely: 1) Anglican Care Center-Hougang; 2) Anglican Care Center-Simei; 3) Anglican Care Center-Bukit Batok; 4) Anglican Care Center-Yishun and 5) Anglican Care Center-Pasir Ris.

1. To investigate the effects of cognitive remediation on:

   * neurocognition (measured by Brief Assessment of Cognition)
   * social cognition (measured by Bell Lysaker Emotion Recognition Task)
   * functional outcomes (Social and Occupational Functioning Assessment Scale and Canadian Occupational Performance Measure).
2. To investigate the mediators for change (eg: motivation and negative symptoms) in cognitive performance and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of schizophrenia or schizoaffective disorder according to Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-V).
* Completed at least ten years of formal education with English as the main instructional language. Participants need to be able to converse in English and understand English instructions, as the cognitive remediation program will be conducted in English.

Exclusion Criteria:

* Known neurological diseases and epilepsy, which affects gains from cognitive remediation.
* Unable to speak and understand English.
* Hospitalized within the past one month.
* Global Assessment of Functioning score of 30 or below, as participants who are too low functioning are unable to benefit from a strategy learning approach.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Brief Assessment of Cognition in Schizophrenia (BACS) | Baseline, post-intervention and 8-week follow-up
  The Brief Assessment of Cognition in Schizophrenia (BACS) assesses the aspects of cognition found to be most impaired and most strongly correlated with outcome in patients with schizophrenia. This assessment was validated and found to be sensitive and highly correlated with the standard battery composite scores in patients (r = 0.76) and healthy controls (r = 0.90) (Keefe et.al., 2004). BACS was also previously normed in English-speaking adult age Singaporeans (Eng et al., 2014), and had demonstrated good convergent validity with education (Lam et al., 2013) and discriminability between healthy controls and schizophrenia (Lam et al., 2014). BACS is now widely used as an outcome measurement for cognitive remediation for schizophrenia.
Bell Lysaker Emotion Recognition Task (BLERT) | Baseline, post-intervention and 8-week follow-up
  The Bell Lysaker Emotion Recognition Task (BLERT) measures the participants' ability to process and recognize seven emotional states: happiness, sadness, fear, disgust, surprise, anger, or no emotion (Bryson, Bell and Lysaker, 1997). The participants will be presented with 21 video clips of an actor demonstrating facial, voice-tonal and upper-body movement cues, while engaging in work-related monologues. Unlike static photos, this measurement appears to simulate real-world situations better and may approximate real world functional outcomes (Pinkham et.al., 2016). Rating was done by computing the total number of correctly recognized emotions (ranging from 0 to 21).
Canadian Occupational Performance Measure (COPM) | Baseline, post-intervention and 8-week follow-up
  The Canadian Occupational Performance Measure (COPM) is a person-centered tool that measures aspects of functional and personal recovery among clients whose occupational performance and participation are affected by their current psychiatric conditions. Through a semi-structured interview, the clients identify activities in self-care, productivity and leisure that are of personal importance and rate their performance and satisfaction in each activity (Law et.al., 1990). Self-perceived performance and satisfaction are rated on a 10-point Likert scale.
Social and Occupational Functioning Assessment Scale (SOFAS) | Baseline, post-intervention and 8-week follow-up
  The Social and Occupational Functioning Assessment Scale (SOFAS) is a global rating of current functioning ranging from 0 to 100, with lower scores representing lower functioning (Goldman et.al., 1992). It differs from GAF scale by focusing on social and occupational functioning independent of the overall severity of the individual's psychological symptoms. SOFAS has been used as a functional outcome measurement in cognitive remediation trials (Au-Yeung et.al., 2023; Harris et.al., 2022; Hodge et.al., 2010).

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Baseline, post-intervention and 8-week follow-up
  This is a 30-item rating instrument, evaluating the presence and severity of positive, negative and general psychopathology of schizophrenia (Kay, Fiszbein & Opler, 1987). The scale was developed from the Brief Psychiatric Rating Scale (BPRS) and the Psychopathology Rating Scale. All 30 items are rated on a 7-point scale (1=absent; 7=extreme). PANSS covers positive and negative symptoms associated with schizophrenia, as well as other symptoms (eg aggression, thought disturbance, depression). Its five-factor model structure has also been validated in the Singapore Schizophrenia Chinese population (Jiang, Sim & Lee, 2013). Hence, the PANSS is a sound instrument to be used for symptom measurement.
Brief Negative Symptom Scale (BNSS) | Baseline, post-intervention and 8-week follow-up
  BNSS consists of five domains of negative symptoms (anhedonia, asociality, avolition, blunted affect, and alogia), which could be clustered into two factors - Motivation-Pleasure (MAP) and Emotional Expressivity (EE) (Kirkpatrick et.al., 2011). A local validation study found that BNSS showed good internal consistency and validity (Ang et.al, 2019). In addition, more severe symptoms as shown in BNSS total, avolition and asociality domains are associated with lower scores on the Global Assessment of Functioning (Ang et.al., 2019).
Brief Regulation of Motivation Scale (BRoMS) | Baseline, post-intervention and 8-week follow-up
  BroMS was initially developed to assess college students' regulation of motivation and two factors were identified: regulation of motivation and willpower (Kim et.al., 2018). Subsequently, a study that adapted and validated it for schizophrenia population found it to be acceptable, feasible and internally consistent, with higher BRoMs scores associated with better work-related skills (Lynch et.al., 2022). The adapted BroMs is a structured interview where participants are told to identify three tasks that they have been working on during the past week. The tasks require participants to maintain their effort over hours or days. The participants are then given 12 statements, where they rate on a 4-point scale, from 'Strongly Disagree' to 'Strongly Agree'. These statements are related to awareness and regulation of motivation.
Weekly Calendar Planning Activity (WCPA) | Baseline, post-intervention and 8-week follow-up
  The Weekly Calendar Planning Activity (WCPA) is a performance-based measure of metacognition, that requires the participant to plan and execute a multiple-step activity. It involves scheduling a list of appointments into a weekly calendar while following rules, avoiding conflicts, monitoring time, and inhibiting distractions, thereby evaluating the participant's planning, error recognition, use of strategies and self-monitoring (Toglia, 2015). Besides scoring for accuracy, the WCPA also scores the difference between the participant's estimated performance and his/her actual performance. Hence, it also evaluates the participant's self-awareness (Kaizerman-Dinerman et.al., 2023).

OTHER OUTCOMES:
The Global Assessment of Functioning Scale (GAF) | Baseline only, to exclude participants with a score of 30 or lower.
  This is carried out prior to recruitment to exclude patients who have a score of 30 or lower. It is a numeric scale (0 through 100) used to rate symptom severity and social, occupational and psychological functioning of adults. The scale is indicated as Axis V in the Diagnostic and Statistical Manual of Mental Disorders-IV-TR and guidelines for scoring have been developed (Aas, 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Bhing-Leet Tan, PhD, Principal Investigator — Bhing-Leet Tan
Locations (5):
- Singapore (5):
  - Anglican Care Center-Bukit Batok, Singapore
  - Anglican Care Center-Hougang, Singapore
  - Anglican Care Center-Pasir Ris, Singapore
  - Anglican Care Center-Simei, Singapore
  - Anglican Care Center-Yishun, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
If the IPD is to be shared eventually, the data to be shared will be the treatment allocation (either experimental or control arm) and the corresponding outcome measurements data.

REFERENCES:
- [Background] Aas IH. Guidelines for rating Global Assessment of Functioning (GAF). Ann Gen Psychiatry. 2011 Jan 20;10:2. doi: 10.1186/1744-859X-10-2. PMID 21251305
- [Background] Au-Yeung C, Bowie CR, Montreuil T, Baer LH, Lecomte T, Joober R, Abdel-Baki A, Jarvis GE, Margolese HC, De Benedictis L, Schmitz N, Thai H, Malla AK, Lepage M. Predictors of treatment attrition of cognitive health interventions in first episode psychosis. Early Interv Psychiatry. 2023 Oct;17(10):984-991. doi: 10.1111/eip.13391. Epub 2023 Jan 18. PMID 36653167
- [Background] Ang MS, Rekhi G, Lee J. Validation of the Brief Negative Symptom Scale and its association with functioning. Schizophr Res. 2019 Jun;208:97-104. doi: 10.1016/j.schres.2019.04.005. Epub 2019 Apr 13. PMID 30987926
- [Background] Eng GK, Lam M, Bong YL, Subramaniam M, Bautista D, Rapisarda A, Kraus M, Lee J, Collinson SL, Chong SA, Keefe RS. Brief assessment of cognition in schizophrenia: normative data in an English-speaking ethnic Chinese sample. Arch Clin Neuropsychol. 2013 Dec;28(8):845-58. doi: 10.1093/arclin/act060. Epub 2013 Aug 1. PMID 23912998
- [Background] Goldman HH, Skodol AE, Lave TR. Revising axis V for DSM-IV: a review of measures of social functioning. Am J Psychiatry. 1992 Sep;149(9):1148-56. doi: 10.1176/ajp.149.9.1148. PMID 1386964
- [Background] Gur RC, Sara R, Hagendoorn M, Marom O, Hughett P, Macy L, Turner T, Bajcsy R, Posner A, Gur RE. A method for obtaining 3-dimensional facial expressions and its standardization for use in neurocognitive studies. J Neurosci Methods. 2002 Apr 15;115(2):137-43. doi: 10.1016/s0165-0270(02)00006-7. PMID 11992665
- [Background] Hancock N, Scanlan JN, Honey A, Bundy AC, O'Shea K. Recovery Assessment Scale - Domains and Stages (RAS-DS): Its feasibility and outcome measurement capacity. Aust N Z J Psychiatry. 2015 Jul;49(7):624-33. doi: 10.1177/0004867414564084. Epub 2014 Dec 19. PMID 25526940
- [Background] Harris AWF, Kightley M, Williams J, Ma C, Dodds C. Does Adding Social Cognitive Remediation Therapy to Neurocognitive Remediation Therapy Improve Outcomes in Young People With a Severe Mental Illness?-The Advantage Trial. Front Psychiatry. 2022 Mar 14;12:789628. doi: 10.3389/fpsyt.2021.789628. eCollection 2021. PMID 35368729
- [Background] Hodge MA, Siciliano D, Withey P, Moss B, Moore G, Judd G, Shores EA, Harris A. A randomized controlled trial of cognitive remediation in schizophrenia. Schizophr Bull. 2010 Mar;36(2):419-27. doi: 10.1093/schbul/sbn102. Epub 2008 Aug 20. PMID 18718884
- [Background] Jiang J, Sim K, Lee J. Validated five-factor model of positive and negative syndrome scale for schizophrenia in Chinese population. Schizophr Res. 2013 Jan;143(1):38-43. doi: 10.1016/j.schres.2012.10.019. Epub 2012 Nov 11. PMID 23148897
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Keefe RS, Goldberg TE, Harvey PD, Gold JM, Poe MP, Coughenour L. The Brief Assessment of Cognition in Schizophrenia: reliability, sensitivity, and comparison with a standard neurocognitive battery. Schizophr Res. 2004 Jun 1;68(2-3):283-97. doi: 10.1016/j.schres.2003.09.011. PMID 15099610
- [Background] Kirkpatrick B, Strauss GP, Nguyen L, Fischer BA, Daniel DG, Cienfuegos A, Marder SR. The brief negative symptom scale: psychometric properties. Schizophr Bull. 2011 Mar;37(2):300-5. doi: 10.1093/schbul/sbq059. Epub 2010 Jun 17. PMID 20558531
- [Background] Lam M, Collinson SL, Eng GK, Rapisarda A, Kraus M, Lee J, Chong SA, Keefe RS. Refining the latent structure of neuropsychological performance in schizophrenia. Psychol Med. 2014 Dec;44(16):3557-70. doi: 10.1017/S0033291714001020. Epub 2014 May 22. PMID 25066336
- [Background] Lam M, Eng GK, Rapisarda A, Subramaniam M, Kraus M, Keefe RSE, Collinson SL. Formulation of the age-education index: measuring age and education effects in neuropsychological performance. Psychol Assess. 2013 Mar;25(1):61-70. doi: 10.1037/a0030548. Epub 2012 Nov 12. PMID 23148648
- [Background] Lynch DA, Brown M, Saperstein A, Stefancic A, Medalia A. Assessing metamotivation in schizophrenia: A pilot study of the Brief Regulation of Motivation Scale (BRoMS). Psychiatry Res. 2022 Nov;317:114799. doi: 10.1016/j.psychres.2022.114799. Epub 2022 Aug 19. PMID 36037743
- [Background] McDonald S, Bornhofen C, Shum D, Long E, Saunders C, Neulinger K. Reliability and validity of The Awareness of Social Inference Test (TASIT): a clinical test of social perception. Disabil Rehabil. 2006 Dec 30;28(24):1529-42. doi: 10.1080/09638280600646185. PMID 17178616
- [Background] Pinkham AE, Harvey PD, Penn DL. Social Cognition Psychometric Evaluation: Results of the Final Validation Study. Schizophr Bull. 2018 Jun 6;44(4):737-748. doi: 10.1093/schbul/sbx117. PMID 28981848
- [Background] Scanlan JN, Hancock N, Honey A. The Recovery Assessment Scale - Domains and Stages (RAS-DS): Sensitivity to change over time and convergent validity with level of unmet need. Psychiatry Res. 2018 Mar;261:560-564. doi: 10.1016/j.psychres.2018.01.042. PMID 29407723
- [Background] Wykes T, Stringer D, Boadu J, Tinch-Taylor R, Csipke E, Cella M, Pickles A, McCrone P, Reeder C, Birchwood M, Fowler D, Greenwood K, Johnson S, Perez J, Ritunnano R, Thompson A, Upthegrove R, Wilson J, Kenny A, Isok I, Joyce EM. Cognitive Remediation Works But How Should We Provide It? An Adaptive Randomized Controlled Trial of Delivery Methods Using a Patient Nominated Recovery Outcome in First-Episode Participants. Schizophr Bull. 2023 May 3;49(3):614-625. doi: 10.1093/schbul/sbac214. PMID 36869733
- [Background] Kim, Y.E., Brady, A.C., Wolters, C.A., 2018. Development and validation of the Brief Regulation of Motivation Scale. Learn. Individ. Differ. 67, 259-265. https://doi.org/ 10.1016/j.lindif.2017.12.010
- [Background] Kiresuk, T. J., Smith, A., & Cardillo, J. E. (2014). Goal attainment scaling: Applications, theory, and measurement. Psychology Press.
- [Background] McDonald, S. (2012) New Frontiers in Neuropsychological Assessment: Assessing Social Perception Using a Standardised Instrument, The Awareness of Social Inference Test. Australian Psychologist 47 (2012) 39-48.
- [Background] Chong NIM, Maniam Y, Chua YC, Tang C. The Implementation and Review of Cognitive Remediation Training for First Episode Psychosis in Singapore. Front Psychiatry. 2021 Nov 30;12:784935. doi: 10.3389/fpsyt.2021.784935. eCollection 2021. PMID 34916979
- [Background] De Mare A, Cantarella M, Galeoto G. Effectiveness of Integrated Neurocognitive Therapy on Cognitive Impairment and Functional Outcome for Schizophrenia Outpatients. Schizophr Res Treatment. 2018 Oct 21;2018:2360697. doi: 10.1155/2018/2360697. eCollection 2018. PMID 30420918
- [Background] Green MF, Kern RS, Braff DL, Mintz J. Neurocognitive deficits and functional outcome in schizophrenia: are we measuring the "right stuff"? Schizophr Bull. 2000;26(1):119-36. doi: 10.1093/oxfordjournals.schbul.a033430. PMID 10755673
- [Background] Hajduk M, Penn DL, Harvey PD, Pinkham AE. Social cognition, neurocognition, symptomatology, functional competences and outcomes in people with schizophrenia - A network analysis perspective. J Psychiatr Res. 2021 Dec;144:8-13. doi: 10.1016/j.jpsychires.2021.09.041. Epub 2021 Sep 24. PMID 34592511
- [Background] McGurk SR, Twamley EW, Sitzer DI, McHugo GJ, Mueser KT. A meta-analysis of cognitive remediation in schizophrenia. Am J Psychiatry. 2007 Dec;164(12):1791-802. doi: 10.1176/appi.ajp.2007.07060906. PMID 18056233
- [Background] Medalia A, Dorn H, Watras-Gans S. Treating problem-solving deficits on an acute care psychiatric inpatient unit. Psychiatry Res. 2000 Dec 4;97(1):79-88. doi: 10.1016/s0165-1781(00)00214-6. PMID 11104859
- [Background] Medalia A, Erlich MD, Soumet-Leman C, Saperstein AM. Translating cognitive behavioral interventions from bench to bedside: The feasibility and acceptability of cognitive remediation in research as compared to clinical settings. Schizophr Res. 2019 Jan;203:49-54. doi: 10.1016/j.schres.2017.07.044. Epub 2017 Jul 30. PMID 28768601
- [Background] Medalia, A., Revheim, N., & Herlands, T. (2009). Cognitive Remediation for Psychological Disorders: Therapist Guide. New York: Oxford University Press.
- [Background] Medalia A, Herlands T, Baginsky C. Rehab rounds: Cognitive remediation in the supportive housing setting. Psychiatr Serv. 2003 Sep;54(9):1219-20. doi: 10.1176/appi.ps.54.9.1219. No abstract available. PMID 12954935
- [Background] Mueller DR, Schmidt SJ, Roder V. One-year randomized controlled trial and follow-up of integrated neurocognitive therapy for schizophrenia outpatients. Schizophr Bull. 2015 May;41(3):604-16. doi: 10.1093/schbul/sbu223. Epub 2015 Feb 22. PMID 25713462
- [Background] Tan BL. Profile of cognitive problems in schizophrenia and implications for vocational functioning. Aust Occup Ther J. 2009 Aug;56(4):220-8. doi: 10.1111/j.1440-1630.2008.00759.x. PMID 20854522
- [Background] Tan BL, Lee SA, Lee J. Social cognitive interventions for people with schizophrenia: A systematic review. Asian J Psychiatr. 2018 Jun;35:115-131. doi: 10.1016/j.ajp.2016.06.013. Epub 2016 Sep 23. PMID 27670776
- [Background] Toglia J (2018) The dynamic interactional model and the multicontext approach. In: Katz N and Toglia J (eds) Cognition, Occupation, and Participation Across the Lifespan. Bethesda, MD: AOTA Press, 355-385.
- [Background] Toglia J, Goverover Y, Johnston MV, Dain B. Application of the Multicontextual Approach in Promoting Learning and Transfer of Strategy Use in an Individual with TBI and Executive Dysfunction. OTJR (Thorofare N J). 2011 Winter;31(1):S53-60. doi: 10.3928/15394492-20101108-09. PMID 24650265
- [Background] Toglia J, Lee A, Steinberg C, Waldman-Levi A. (2020) Establishing and measuring treatment fidelity of a complex cognitive rehabilitation intervention: The multicontext approach. British Journal of Occupational Therapy. 83(6):363-374. doi:10.1177/0308022619898091
- [Background] Ventura J, Hellemann GS, Thames AD, Koellner V, Nuechterlein KH. Symptoms as mediators of the relationship between neurocognition and functional outcome in schizophrenia: a meta-analysis. Schizophr Res. 2009 Sep;113(2-3):189-99. doi: 10.1016/j.schres.2009.03.035. Epub 2009 Jul 22. PMID 19628375
- [Background] Wykes T, Huddy V, Cellard C, McGurk SR, Czobor P. A meta-analysis of cognitive remediation for schizophrenia: methodology and effect sizes. Am J Psychiatry. 2011 May;168(5):472-85. doi: 10.1176/appi.ajp.2010.10060855. Epub 2011 Mar 15. PMID 21406461
- [Background] Bryson G, Bell M, Lysaker P. Affect recognition in schizophrenia: a function of global impairment or a specific cognitive deficit. Psychiatry Res. 1997 Jul 4;71(2):105-13. doi: 10.1016/s0165-1781(97)00050-4. PMID 9255855
- [Background] Law M, Baptiste S, McColl M, Opzoomer A, Polatajko H, Pollock N. The Canadian occupational performance measure: an outcome measure for occupational therapy. Can J Occup Ther. 1990 Apr;57(2):82-7. doi: 10.1177/000841749005700207. PMID 10104738
- [Background] Toglia J. Weekly calendar planning activity: a performance test of executive function. AOTA Press; 2015.
- [Background] Kaizerman-Dinerman A, Roe D, Demeter N, Josman N. Do symptoms moderate the association between participation and executive functions outcomes among people with schizophrenia? BMC Psychiatry. 2023 Jan 17;23(1):42. doi: 10.1186/s12888-022-04510-0. PMID 36650458
- [Derived] Tan BL, Tan N, Koh V, Poh L, Medalia A. Integrative Neuro-social cognitive Strategy Programme for Instilling REcovery (INSPIRE): a community-based cognitive remediation trial-study procotol. BMC Psychiatry. 2024 Sep 19;24(1):621. doi: 10.1186/s12888-024-06070-x. PMID 39300363